CLINICAL TRIAL: NCT02832999
Title: Short Term Effect of Liraglutide Versus Vildagliptine on Insulin Secretion and Insulin Sensitivity in a Sub Saharan African Population With Type 2 Diabetes
Brief Title: Short Term Effect of Liraglutide Versus Vildagliptine on Insulin Secretion and Insulin Sensitivity in Type 2 Diabetes
Acronym: LIRAVIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: University of Yaounde 1 (Other); University of Buea (Other)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor of Endocrinology and Diabetes, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNO20163
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; GLP-1; Insulin secretion; insulin sensitivity; Africa; Liraglutide; Vildaglipin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Liraglutide; Vildagliptin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sub cutaneous liraglutide (Experimental): once daily add-on subcutaneous injection of Liraglutide at 0.6mg/day for 1 week increased to 1.2mg the second week
  Interventions: Drug: sub cutaneous liraglutide
- Oral Vildagliptin (Active Comparator): Once daily oral 100mg of Vildagliptine for two weeks
  Interventions: Drug: Oral Vildagliptin

INTERVENTIONS:
Drug: sub cutaneous liraglutide — Liraglutide 1.2mg/day
  Other Names: Victoza
  Arms: sub cutaneous liraglutide
Drug: Oral Vildagliptin — Vildagliptin 50mg/day
  Other Names: Galvus
  Arms: Oral Vildagliptin

SUMMARY:
This is a single blind randomised controlled clinical trial in uncontrolled type 2 Diabetes mellitus patients on oral glucose lowering agents, and naive to incretinomimetic. Participants will be randomised in two Arms : arm 1 receiving Liraglutide at 1,2 mg/day and arm 2 Vildagliptine at 100mg/day over 14 days. The two arms will be compared for 14-day changes in insulin secretion and insulin sensitivity.

DETAILED DESCRIPTION:
Incretinomimetics include exogenous Glucagon-Like Peptide analogs (GLP1a) such as Liraglutide, and inhibitors of Dipeptidyl peptidase IV (DPP4i) that prolong the half-life of endogenous GLP1 such as Vildagliptin. It remains unclear which of the two strategies (exogenous GLP1 or prolonging half-life of endogenous GLP1) have better short term effect on insulin sensitivity and insulin secretion in people living with type 2 diabetes.

This study aims to investigate the short-term metabolic effects of a GLP-1 analog Liraglutide versus a DPP4i Vildagliptin. It is a randomized, controlled, single-blinded clinical trial. Study population consists of uncontrolled type 2 diabetes mellitus patients (HbA1c≥7%) under mono or bi oral anti-diabetic therapy, naïve of any incretinomimetic treatment. Participants are randomized in 2 arms. The intervention in arm 1 consists of add-on subcutaneous Liraglutide at 0.6mg/day for 1 week increased to 1.2mg the second week. In the second arm, it consists of oral Vildagliptine at 100mg daily for two weeks. The primary outcome is the variation in euglycaemic hyperinsulinaemic clamp-derived insulin sensitivity before randomization and the day after intervention, secondary outcomes include 14-day changes in insulin secretion during a mixed meal tolarance test, body weight and body composition, and an indirect calorimetry measured resting energy expenditure. Changes from baseline to 14 days in serum creatinine and alanine amino transferase, C-reactive protein and lipid profile will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus known for at least one year
* Uncontrolled glycaemic profile with HbA1c ≥ 7% on oral antidiabetic mono or bi-therapy
* Naïve of incretinomimetic treatment
* Informed consent

Exclusion Criteria:

* Change in antidiabetic treatment less than 3 months prior to inclusion
* Pancreatitis
* Alanine amino transferase > 3 times the normal values
* Pregnant or breastfeeding women
* Estimated glomerular filtration rate < 60ml/min
* Infection less than 10 days prior to inclusion or during the study
* Acute complication of diabetes
* Total haemoglobin < 11g/dL in women or < 13g/dL in men
* Withdrawal of consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Insulin sentivity | 2 weeks
  2-week change in clamp-measured insulin sensitivity

SECONDARY OUTCOMES:
insulin secretion | 2 weeks
  2-week change in meal test measured insulin secretion
lipid profile | 2 weeks
  2-week change in fasting serum lipids
body weight | 2 weeks
  2-week change in body weight

OTHER OUTCOMES:
Renal function | 2 weeks
  2-week change in serum creatinine
Inflammation | 2 weeks
  2-week change in C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Eugène Sobngwi, Principal Investigator — Yaounde Central Hospital
Locations (1):
- National Obesity Centre, Yaoundé, Cameroon